CLINICAL TRIAL: NCT05894902
Title: Open-Label Dose-Ranging Study of Oral SM-001 in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Advanced Integrative Medical Science Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SM-001
Record Dates: First submitted 2023-03-15; First posted 2023-06-08 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Major Depression; Post Traumatic Stress Disorder
Keywords: Banisteriopsis caapi; Psychotria viridis; ayahuasca; ethnomedicine; N,N-dimethyltryptamine (DMT); harmine (HAR); harmaline; tetrahydroharmine
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Subjects will be consecutively accrued to one of three study groups, starting at the lowest dose, Level 1 ("low" dose), and proceeding to the next higher dose level. Each subject will receive one dose of the Study Drug orally at the Clinical Study Site, according to their assigned dose Level. Dose levels vary by volume:
  Level 1: 0.5 mL/kg ("low"; 50% of usual dose) N=4 (2M/2F) Level 2: 1 ml/kg ("medium"; 100% of usual dose) N=4 (2M/2F) Level 3: 2 ml/kg ("high"; 200% of usual dose) N=4 (2M/2F)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open label Phase I safety & dose finding study: low dose group (Active Comparator): 4 study participants will receive a low oral dose (0.5 mL/Kg) of SM-001
  Interventions: Drug: SM-001
- Open label Phase I safety & dose finding study: medium dose group (Active Comparator): 4 study participants will receive a medium oral dose (1.0 mL/Kg) of SM-001
  Interventions: Drug: SM-001
- Open label Phase I safety & dose finding study: high dose group (Active Comparator): 4 study participants will receive a high oral dose (2.0 mL/Kg) of SM-001
  Interventions: Drug: SM-001

INTERVENTIONS:
Drug: SM-001 — The Investigational New Drug SM-001 is formulated as a hot water decoction of two proprietary clonal cultivars of the Peruvian plants, Banisteriopsis caapi (BC) and Psychotria viridis (PV).
  Other Names: Ayahuasca

SUMMARY:
Phase I safety and dose finding study of a standardized Ayahuasca analog (SM-001) in healthy adult volunteers

DETAILED DESCRIPTION:
The Investigational New Drug SM-001 is formulated as a hot water decoction of two clonal cultivars of the Peruvian plants, Banisteriopsis caapi (BC) and Psychotria viridis (PV). It represents a modern formulation of an ancient Amazonian botanical medicine, "ayahuasca" ("vine of the soul") that is used by many native South American indigenous and mestizo groups for both religious and medicinal purposes.

This initial Phase 1 study is to be conducted as an open label, dose-ranging safety assessment of a single dose of SM-001 taken orally by healthy adult volunteers. Twelve adult men and women, ages 25-65 years, will be consecutively assigned to one of three dose levels, 4 subjects per group (2 M; 2 F). In the presence of the Clinical Investigator(s), each subject will receive a single dose of SM-001, administered at the Clinical Study Site as a liquid at one of three dose levels: 0.25, 0.5, or1.5 ml SM-001 per kg body weight. To assess systemic exposure to SM-001, plasma levels of the four biomarkers, dimethyltryptamine, harmine, tetrahydroharmine, and harmaline will be measured. Blood samples will be drawn at baseline, HR 0 (pre-Study Drug dose), and then at HR 1, 2, 4, 8, and 24 post dose. Subjects will return to the Clinical Study Site at Study Day 28 for a final in-person assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults: men and women ages 25-65 years of age
* Previous experience with a psychedelic drug
* Vital Signs within normal limits for temperature (oral), respiratory rate, heart rate
* Normal blood pressure (for age) in the absence of antihypertensive drugs
* Normal complete blood count and differential, platelets, coagulation ((PT/PTT)
* Liver function tests ≤ 1.5X upper limits of normal
* Renal function (BUN, serum Creatinine) - within normal limits
* Able to understand and willing to comply with Study Protocol requirements.
* Willing to abstain from alcohol for at least 72 hours prior to and following Study Day 0
* No use of recreational drugs for at least 14 days prior to Study Day 0.
* Women who are not pregnant or lactating.

Exclusion Criteria (None can apply):

* Body Mass Index > 30 or < 20
* Systemic condition that includes, but is not limited to: hematological, immunological, hepatic, renal, cardiac, neurological conditions that is under current treatment or causes abnormal physical or laboratory parameters.
* History of seizures
* History of drug or alcohol abuse
* History of psychiatric disorder or history of significant trauma, as defined by DSM- V.
* Use of SSRIs, MAO inhibitors, or other psychoactive compounds either pharmaceutical drugs or botanical in origin (i.e., 5-HTP, St John's Wort)
* Any condition which, in the opinion of the Investigators, would preclude the use of the test article or the successful completion of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 1-28 days
  To evaluate safety and tolerability of SM-001 in healthy adults following a single oral dose, at one of three different dose levels. The Incidence of Treatment-Emergent Adverse Events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE).
  Percentage of participants with at least one safety event [Time Frame: Baseline up to Day 28 ] Safety will be evaluated by the monitoring of adverse events (AEs), vital signs, blood pressure, heart rate, pulse oximetry, electrocardiogram (ECG) evaluations, clinical laboratory assessments and physical examination findings.

SECONDARY OUTCOMES:
Short-term psychological impact | 24 hours after single drug session
  To assess short-term psychological impact of a single dose of SM-001 at three different dose levels in healthy adults by asking each study subject to complete a questionnaire called the Hallucinogenic Rating Scale 24 hours after the single experimental drug session. This is an 85 item questionnaire with each item rated 0-4 with a maximum score of 340. A higher score correlates with a more intense psychological experience.
Longer-term psychological impact | Day 7 after a single drug session
  To assess longer-term psychological impact of a single dose of SM-001 at three different dose levels in healthy adults by asking each study subject to complete a questionnaire called the Persisting Effects Questionnaire 7 days following the single experimental drug session.
  The Persisting Effects Questionnaire includes 140 of the items that are rated on a 6-point scale (0=none, not at all; 1=so slight cannot decide; 2=slight; 3=moderate; 4=strong; 5=extreme, more than ever before in your life and stronger than 4).
Bioavailability of SM-001 | Day 1-2
  To determine the blood, urine and feces levels of plant alkaloids including dimethyltryptamine, harmine, tetrahydroharmine and harmaline in ng/mL following a single oral dose of SM-001.
Effects of a single dose of SM-001 on blood levels of brain derived nerve growth factor | Day 1-28
  Brain Derived Neurotrophic Factor will be quantitated (ng/mL) is each study subject's blood on the day before and the day after the SM-001 drug session.
Effects of a single dose of SM-001 on blood cortisol blood levels | Day 1 - 28
  Cortisol levels in each study subject's blood will be measured (mg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Leanna J Standish, ND PhD, Principal Investigator — AIMS Institute
Locations (1):
- AIMS Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarons DH, Rossi GV, Orzechowski RF. Cardiovascular actions of three harmala alkaloids: harmine, harmaline, and harmalol. J Pharm Sci. 1977 Sep;66(9):1244-8. doi: 10.1002/jps.2600660910. PMID 903860
- [Background] Barrett FS, Johnson MW, Griffiths RR. Validation of the revised Mystical Experience Questionnaire in experimental sessions with psilocybin. J Psychopharmacol. 2015 Nov;29(11):1182-90. doi: 10.1177/0269881115609019. Epub 2015 Oct 6. PMID 26442957
- [Background] Brown CS, Bryant SG. Monoamine oxidase inhibitors: safety and efficacy issues. Drug Intell Clin Pharm. 1988 Mar;22(3):232-5. doi: 10.1177/106002808802200311. PMID 3284731
- [Background] Hamill J, Hallak J, Dursun SM, Baker G. Ayahuasca: Psychological and Physiologic Effects, Pharmacology and Potential Uses in Addiction and Mental Illness. Curr Neuropharmacol. 2019;17(2):108-128. doi: 10.2174/1570159X16666180125095902. PMID 29366418
- [Background] Callaway JC, Raymon LP, Hearn WL, McKenna DJ, Grob CS, Brito GS, Mash DC. Quantitation of N,N-dimethyltryptamine and harmala alkaloids in human plasma after oral dosing with ayahuasca. J Anal Toxicol. 1996 Oct;20(6):492-7. doi: 10.1093/jat/20.6.492. PMID 8889686
- [Background] Da Prada M, Zurcher G, Wuthrich I, Haefely WE. On tyramine, food, beverages and the reversible MAO inhibitor moclobemide. J Neural Transm Suppl. 1988;26:31-56. PMID 3283290
- [Background] dos Santos RG. Safety and side effects of ayahuasca in humans--an overview focusing on developmental toxicology. J Psychoactive Drugs. 2013 Jan-Mar;45(1):68-78. doi: 10.1080/02791072.2013.763564. PMID 23662333
- [Background] Dos Santos RG, Grasa E, Valle M, Ballester MR, Bouso JC, Nomdedeu JF, Homs R, Barbanoj MJ, Riba J. Pharmacology of ayahuasca administered in two repeated doses. Psychopharmacology (Berl). 2012 Feb;219(4):1039-53. doi: 10.1007/s00213-011-2434-x. Epub 2011 Aug 13. PMID 21842159
- [Background] Santos RG, Landeira-Fernandez J, Strassman RJ, Motta V, Cruz AP. Effects of ayahuasca on psychometric measures of anxiety, panic-like and hopelessness in Santo Daime members. J Ethnopharmacol. 2007 Jul 25;112(3):507-13. doi: 10.1016/j.jep.2007.04.012. Epub 2007 Apr 25. PMID 17532158
- [Background] Dominguez-Clave E, Soler J, Elices M, Pascual JC, Alvarez E, de la Fuente Revenga M, Friedlander P, Feilding A, Riba J. Ayahuasca: Pharmacology, neuroscience and therapeutic potential. Brain Res Bull. 2016 Sep;126(Pt 1):89-101. doi: 10.1016/j.brainresbull.2016.03.002. Epub 2016 Mar 11. PMID 26976063
- [Background] Gable RS. Risk assessment of ritual use of oral dimethyltryptamine (DMT) and harmala alkaloids. Addiction. 2007 Jan;102(1):24-34. doi: 10.1111/j.1360-0443.2006.01652.x. PMID 17207120
- [Background] Gillin JC, Tinklenberg J, Stoff DM, Stillman R, Shortlidge JS, Wyatt RJ. 5-Methoxy-N,N-dimethyltryptamine: behavioral and toxicological effects in animals. Biol Psychiatry. 1976 Jun;11(3):355-8. No abstract available. PMID 820383
- [Background] Griffiths R, Richards W, Johnson M, McCann U, Jesse R. Mystical-type experiences occasioned by psilocybin mediate the attribution of personal meaning and spiritual significance 14 months later. J Psychopharmacol. 2008 Aug;22(6):621-32. doi: 10.1177/0269881108094300. Epub 2008 Jul 1. PMID 18593735
- [Background] Grob CS, McKenna DJ, Callaway JC, Brito GS, Neves ES, Oberlaender G, Saide OL, Labigalini E, Tacla C, Miranda CT, Strassman RJ, Boone KB. Human psychopharmacology of hoasca, a plant hallucinogen used in ritual context in Brazil. J Nerv Ment Dis. 1996 Feb;184(2):86-94. doi: 10.1097/00005053-199602000-00004. PMID 8596116
- [Background] Kamel SH, Ibrahim TM, Hamza SM. Effect of harmine and harmaline hydrochloride on pregnancy in white rats. Zentralbl Veterinarmed A. 1971 May;18(3):230-3. doi: 10.1111/j.1439-0442.1971.tb00573.x. No abstract available. PMID 4997511
- [Background] Luna LE. The healing practices of a Peruvian shaman. J Ethnopharmacol. 1984 Jul;11(2):123-33. doi: 10.1016/0378-8741(84)90035-7. PMID 6387284
- [Background] Marwood JF, Huston V, Wall KT. Some cardiovascular effects of monoamine oxidase inhibitors in unanaesthetized rats. Clin Exp Pharmacol Physiol. 1985 Mar-Apr;12(2):161-8. doi: 10.1111/j.1440-1681.1985.tb02319.x. PMID 3839173
- [Background] McCabe BJ. Dietary tyramine and other pressor amines in MAOI regimens: a review. J Am Diet Assoc. 1986 Aug;86(8):1059-64. PMID 3525654
- [Background] McKenna DJ. Ayahuasca and human destiny. J Psychoactive Drugs. 2005 Jun;37(2):231-4. doi: 10.1080/02791072.2005.10399805. PMID 16149337
- [Background] McKenna DJ, Towers GH, Abbott F. Monoamine oxidase inhibitors in South American hallucinogenic plants: tryptamine and beta-carboline constituents of ayahuasca. J Ethnopharmacol. 1984 Apr;10(2):195-223. doi: 10.1016/0378-8741(84)90003-5. PMID 6587171
- [Background] Naranjo P. Hallucinogenic plant use and related indigenous belief systems in the Ecuadorian Amazon. J Ethnopharmacol. 1979 Apr;1(2):121-45. doi: 10.1016/0378-8741(79)90003-5. PMID 542010
- [Background] O'Hearn E, Molliver ME. Degeneration of Purkinje cells in parasagittal zones of the cerebellar vermis after treatment with ibogaine or harmaline. Neuroscience. 1993 Jul;55(2):303-10. doi: 10.1016/0306-4522(93)90500-f. PMID 8377927
- [Background] Oliveira CD, Moreira CQ, de Sa LR, Spinosa Hde S, Yonamine M. Maternal and developmental toxicity of ayahuasca in Wistar rats. Birth Defects Res B Dev Reprod Toxicol. 2010 Jun;89(3):207-12. doi: 10.1002/bdrb.20244. PMID 20549682
- [Background] Palhano-Fontes F, Andrade KC, Tofoli LF, Santos AC, Crippa JA, Hallak JE, Ribeiro S, de Araujo DB. The psychedelic state induced by ayahuasca modulates the activity and connectivity of the default mode network. PLoS One. 2015 Feb 18;10(2):e0118143. doi: 10.1371/journal.pone.0118143. eCollection 2015. PMID 25693169
- [Background] Pic-Taylor A, da Motta LG, de Morais JA, Junior WM, Santos Ade F, Campos LA, Mortari MR, von Zuben MV, Caldas ED. Behavioural and neurotoxic effects of ayahuasca infusion (Banisteriopsis caapi and Psychotria viridis) in female Wistar rat. Behav Processes. 2015 Sep;118:102-10. doi: 10.1016/j.beproc.2015.05.004. Epub 2015 Jun 3. PMID 26049017
- [Background] Pitol DL, Siessere S, Dos Santos RG, Rosa ML, Hallak JE, Scalize PH, Pereira BF, Iyomasa MM, Semprini M, Riba J, Regalo SC. Ayahuasca Alters Structural Parameters of the Rat Aorta. J Cardiovasc Pharmacol. 2015 Jul;66(1):58-62. doi: 10.1097/FJC.0000000000000243. PMID 25714595
- [Background] Riba J, McIlhenny EH, Valle M, Bouso JC, Barker SA. Metabolism and disposition of N,N-dimethyltryptamine and harmala alkaloids after oral administration of ayahuasca. Drug Test Anal. 2012 Jul-Aug;4(7-8):610-6. doi: 10.1002/dta.1344. Epub 2012 Apr 19. PMID 22514127
- [Background] Riba J, Rodriguez-Fornells A, Strassman RJ, Barbanoj MJ. Psychometric assessment of the Hallucinogen Rating Scale. Drug Alcohol Depend. 2001 May 1;62(3):215-23. doi: 10.1016/s0376-8716(00)00175-7. PMID 11295326
- [Background] Kiraga MK, Mason NL, Uthaug MV, van Oorsouw KIM, Toennes SW, Ramaekers JG, Kuypers KPC. Persisting Effects of Ayahuasca on Empathy, Creative Thinking, Decentering, Personality, and Well-Being. Front Pharmacol. 2021 Oct 1;12:721537. doi: 10.3389/fphar.2021.721537. eCollection 2021. PMID 34658861
- [Background] Cameron LP, Benson CJ, Dunlap LE, Olson DE. Effects of N, N-Dimethyltryptamine on Rat Behaviors Relevant to Anxiety and Depression. ACS Chem Neurosci. 2018 Jul 18;9(7):1582-1590. doi: 10.1021/acschemneuro.8b00134. Epub 2018 Apr 24. PMID 29664276
- [Background] Sklerov J, Levine B, Moore KA, King T, Fowler D. A fatal intoxication following the ingestion of 5-methoxy-N,N-dimethyltryptamine in an ayahuasca preparation. J Anal Toxicol. 2005 Nov-Dec;29(8):838-41. doi: 10.1093/jat/29.8.838. PMID 16356341
- [Background] Strassman RJ, Qualls CR, Uhlenhuth EH, Kellner R. Dose-response study of N,N-dimethyltryptamine in humans. II. Subjective effects and preliminary results of a new rating scale. Arch Gen Psychiatry. 1994 Feb;51(2):98-108. doi: 10.1001/archpsyc.1994.03950020022002. PMID 8297217
- [Background] Bilhimer MH, Schult RF, Higgs KV, Wiegand TJ, Gorodetsky RM, Acquisto NM. Acute Intoxication following Dimethyltryptamine Ingestion. Case Rep Emerg Med. 2018 Feb 27;2018:3452691. doi: 10.1155/2018/3452691. eCollection 2018. PMID 29682363
- [Background] Wehner FC, Thiel PG, van Rensburg SJ. Mutagenicity of alkaloids in the Salmonella/microsome system. Mutat Res. 1979 Feb;66(2):187-90. doi: 10.1016/0165-1218(79)90065-x. No abstract available. PMID 372800
- [Background] Wiltshire PE, Hawksworth DL, Edwards KJ. Light microscopy can reveal the consumption of a mixture of psychotropic plant and fungal material in suspicious death. J Forensic Leg Med. 2015 Aug;34:73-80. doi: 10.1016/j.jflm.2015.05.010. Epub 2015 Jun 4. PMID 26165663
- [Background] Yritia M, Riba J, Ortuno J, Ramirez A, Castillo A, Alfaro Y, de la Torre R, Barbanoj MJ. Determination of N,N-dimethyltryptamine and beta-carboline alkaloids in human plasma following oral administration of Ayahuasca. J Chromatogr B Analyt Technol Biomed Life Sci. 2002 Nov 5;779(2):271-81. doi: 10.1016/s1570-0232(02)00397-5. PMID 12361741